CLINICAL TRIAL: NCT06386731
Title: Continuous Versus Intermittent Phototherapy in Treatment of Neonatal Jaundice: A Randomized Controlled Trial
Brief Title: Continuous Versus Intermittent Phototherapy in Treatment of Neonatal Jaundice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Sibel Sevuk Ozumut, pediatric clinic chief assistant, MD, Goztepe Prof Dr Suleyman Yalcın City Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYNEO-01
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Neonatal Jaundice; Phototherapy Complication
Keywords: indirect hyperbilirubinemia; continuous phototherapy; intermittent phototherapy; phototherapy side effects
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Intervention Model Description: This was a single-center, with block randomisation [1:1], open-label, parallel group study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intermittent phototherapy group (Active Comparator): In the intermittent phototherapy group, phototherapy will be applied for 1 hour, phototherapy will be turned off for 2 hours, and time will be left for cleansing from the skin. The 3-hour cycle is completed twice and the 6-hour session is completed, and at the end, the total bilirubin will be measured and the hourly bilirubin decrease rate will be calculated.
  Interventions: Other: Intermittent Phototherapy
- continuous phototherapy group (Other): In the continuous phototherapy group, total bilirubin will be measured at the end of 6 hours of uninterrupted phototherapy and the hourly bilirubin decrease rate will be calculated.
  Interventions: Other: Intermittent Phototherapy

INTERVENTIONS:
Other: Intermittent Phototherapy — 2-hour phototherapy application in the intervention group
  Other Names: Phototherapy duration

SUMMARY:
One of the most common diseases in the neonatal period is indirect hyperbilirubinemia (IHB). After phototherapy was discovered accidentally in 1958, it has been used as the most effective treatment method for IHD for more than 60 years. Sources that provide phototherapy are developing rapidly technologically. However, there is no clearly defined usage table in the literature for applying phototherapy with faster effects and fewer side effects. In recent years, the use of intermittent phototherapy has been recommended with similar effectiveness. Phototherapy has significant side effects such as dehydration, diarrhea, chromosome breaks, retinal damage, skin rashes, hypocalcemia, thrombocytopenia. As phototherapy exposure decreases, its side effects decrease.In our study; We plan to find the most ideal method in the treatment of IHB by comparing intermittent PT with continuous phototherapy in terms of effectiveness. We aim to achieve the best bilirubin reduction and minimal side effects with less exposure to phototherapy.

DETAILED DESCRIPTION:
n the intermittent phototherapy group, phototherapy will be applied for 1 hour and phototherapy will be turned off for 2 hours, allowing time for the skin to be cleaned. The 3-hour cycle is completed twice and the 6-hour session is completed, and at the end, the total bilirubin will be measured and the hourly bilirubin decrease rate will be calculated.

In the continuous phototherapy group, total bilirubin will be measured at the end of 6 hours of uninterrupted phototherapy and the hourly bilirubin decrease rate will be calculated.

It was planned to compare the effectiveness of the two groups in terms of the bilirubin level reduced as a result of 6-hour sessions, hourly reduction rate, rebound bilirubin level, total phototherapy time received, hospitalization time, and additional treatments required.

It was planned to compare both groups in terms of the frequency of side effects such as the number of defecations, body temperature changes, and skin rash during the phototherapy session.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria was being a late preterm or term neonate who had IHB in the first 15 days of life-

Exclusion Criteria:

* Those who had sTB values at the blood exchange limit according to the nomogram, any associated congenital anomalies including chromosomal anomalies or were less than 34th gestational week were excluded.

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 225 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Comparison of the effectiveness of CPT and IPT | 10 months
  The primary outcome was to compare the therapeutic efficacy of IPT and CPT

SECONDARY OUTCOMES:
Comparison of side effect frequency of CPT and IPT | 10 months
  Comparison of frequency of skin rash, increase in body temperature, diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Fahri Ovalı, Prof, Study Chair — İstanbul medeniyet University
Locations (1):
- Göztepe Prof. Dr. Suleyman Yalcin City Hopital, Kadıköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years
Access Criteria: Medical doctors and medical students who will conduct research on the subject can access the data.

REFERENCES:
- See also: Intermittent versus continuous phototherapy for the treatment of neonatal non-hemolytic moderate hyperbilirubinemia in infants more than 34 weeks of gestational age: a randomized controlled trial. — https://doi.org/10.1007/s00431-014-2373-8
- See also: Comparison of efficacy, safety & satisfaction of intermittent versus continuous phototherapy in hyperbilirubinaemic newborns ≥35 week gestation: A randomized controlled trial. — https://doi.org/10.4103/ijmr.IJMR_2156_18
- See also: Sixty years of phototherapy for neonatal jaundice - from serendipitous observation to standardized treatment and rescue for millions — https://doi.org/10.1038/s41372-019-0439-1